CLINICAL TRIAL: NCT01341860
Title: Investigation of Genetic Marker Associated With Obesity in Koreans, A Single-nucleotide Polymorphism(SNP) Analysis for Korean Obese
Brief Title: Investigation of Genetic Marker Associated With Obesity in Koreans
Acronym: IGM-OK
Status: Terminated | Type: Observational
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Jae-Young Um, Kyung Hee University
Other Study IDs: KHU-110421; KHU-1101 (Other Grant/Funding Number: Kyung Hee University)
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- controls: control group with a BMI of less thatn 25kg/m2
- obese group: Obese patients with BMI 25-30 kg/m2

SUMMARY:
A single-nucleotide polymorphism (SNP) analysis of DNA obtained from peripheral blood of the obese patients and the normal control will be performed to find genetic marker for obesity

ELIGIBILITY:
Inclusion Criteria:

* BMI 25~30kg/m2

Exclusion Criteria:

* All were nonsmokers and had no evidence of cancer, liver, renal, hematological disease or other metabolic disorders other than obesity

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: obese patients with BMI 25~30 kg/m2 who visited Kyung Hee University Hospital, Seoul, Korea
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2000-01; Primary Completion 2003-12 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
genotyping for the SNP associated with BMI | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Young Um, PhD, Principal Investigator — Kyunghee University